CLINICAL TRIAL: NCT00293150
Title: Determine the Effectiveness of Eplerenone in Reversing Diastolic Dysfunction, Improving Endothelial Function, and Suppressing Natriuretic Peptides and Collagen Turnover in Patients With Diastolic Heart Failure ( PREDICT Study)
Brief Title: Reversing Endothelial and Diastolic Dysfunction and Improving Collagen Turnover in Diastolic Heart Failure
Acronym: PREDICT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of eligible patients
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6242
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diastolic Heart Failure
Keywords: diastolic heart failure; heart failure
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind placebo vs eplerenone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eplerenone (Active Comparator): Eplerenone 25mg daily for 2 weeks Titrated to Eplerenone 50mg daily
  Interventions: Drug: Eplerenone
- Placebo (Placebo Comparator): Placebo dosed daily
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone
  Other Names: Inspra

SUMMARY:
The principle aim is to determine the efficacy of eplerenone in patients with diastolic heart failure to reverse cardiac remodeling and to improve diastolic function.

DETAILED DESCRIPTION:
The study will be a single center, double-blind, randomized, parallel group trial enrolling a minimum of 80 patients designed to determine the efficacy of eplerenone in subjects with diastolic heart failure. Prior to administration of study medication, a medical history, physical exam, blood draw, electrocardiogram, 2D echocardiogram, and cardiomyopathy questionnaire will be performed. Subjects will then be randomized to receive either eplerenone 25 mg once daily or placebo for 2 weeks. At the Week 2 visit all patients will be titrated up to the next dose (50 mg eplerenone once daily or placebo). Each study arm will have 40 subjects who will participate for 9 months. Follow-up assessments will be completed at 1 week, 2 weeks, 1 month, 3 months, 6 months, and 9 months.

Starting at the Month 1 visit, any subjects with uncontrolled blood pressure will be administered add-on therapy of HCTZ (starting dose of 12.5 mg daily, that may titrate up to 25 mg daily) and/or amlodipine (starting dose at 5 mg daily, that may titrate up to 10 mg daily). Any subject who receives add-on therapy must have their blood pressure checked within 2 weeks. Uncontrolled blood pressure may be treated by either increasing the add-on therapy dose or increasing the add-on therapy regimen to include both add-on drugs. Changes in add-on therapy require blood pressure checks within 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Male or non-pregnant female (if female, either post-menopausal, or if of child-bearing potential, using adequate contraception e.g. hormonal or barrier methods, or surgically sterile, and not lactating)
2. Age >/= 18 years of age
3. Present or prior history of symptoms of heart failure (dyspnea, fatigue) consistent with diagnosis of diastolic heart failure, following optimized medical therapy including blood pressure control with ACE inhibitors and/or beta-blockers for 2 weeks or over.
4. Echocardiographic evidence of preserved left ventricular systolic function (LVEF >/= 45%) and evidence of diastolic dysfunction (by transmitral inflow, pulmonary venous flow, color M-mode and/or tissue Doppler).
5. Signed informed consent

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

1. Unwilling to participate for the 9-month duration of the study
2. Significant primary valvular, pulmonary or congenital cardiac disease believed to be the cause of dyspnea
3. Life expectancy or planned cardiac transplantation <9 months
4. History of hypertrophic obstructive cardiomyopathy
5. Unstable angina or ischemia requiring revascularization
6. Renal insufficiency (Cr >2.0 mg/dL in males and >1.8 mg/dl in females, or modified Cockcroft-Gault estimate of creatinine clearance <30 mL/min) at enrollment
7. Known hypersensitivity to spironolactone or eplerenone
8. Decompensated heart failure or clinical evidence of instability at the time of enrollment 9 History of hyperkalemia (>6.0 mg/dL) with spironolactone

10. Use of spironolactone or amiloride within 30 days 11. Poorly controlled seating blood pressure at the time of drug initiation:

* Systolic blood pressure >160 mmHg; and/or
* Diastolic blood pressure >100 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of eplerenone | 9 months
  Improved diastolic function

SECONDARY OUTCOMES:
Degree of change | 9 months
  degree of changes in natriuretic peptide production, endothelial function and collagen turnover

CONTACTS AND LOCATIONS:
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No